CLINICAL TRIAL: NCT00005746
Title: Community Site Coronary Risk Control in Black Families
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5012; R01HL058625 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Coronary Heart Disease Risk Reduction
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease

SUMMARY:
To test the effectiveness of a community site neighborhood health worker/nurse (NHW/N) case management strategy for coronary heart disease risk reduction compared with usual care in apparently healthy African American siblings of persons with documented premature coronary heart disease.

DETAILED DESCRIPTION:
BACKGROUND:

The rationale for this program proceeded from the markedly increased risk of initial coronary events in siblings with coronary artery disease with onset before age 50. There is an excess of treatable coronary heart disease risk factors in such siblings and a high prevalence of adult atherosclerosis.

DESIGN NARRATIVE:

The study recruited 364 siblings of individuals with early coronary disease. Eligible subjects were randomized to community-based care (CBC) or enhanced primary care (EPC) with a community health site neighborhood health worker/nurse for 1 year follow up. Intervention participants were stratified based on results of treadmill testing to either more or less aggressive management of their lipids according to National Cholesterol Education Program guidelines. All positive participants on the exercise stress test were directly referred to their physicians. Diabetics were referred to their primary physician for treatment. Intervention in the intervention group was carried out on traditional coronary heart disease (CHD) risk factors including diet, physical activity, blood pressure, LDL cholesterol, and cigarette smoking. The intervention built on a prior sibling study in Blacks and whites.

The approach was that, rather than carrying out the intervention at the central John Hopkins Clinic, thus requiring transportation of potentially anxious participants to a strange environment, the new interventions were carried out by trained local NHWs in a more accessible local community site. The nutrition interventions used fat counters that focused on total fat gram goals, and intervention was carried out by the NHW/N with assistance from cookbooks appropriate for African American households. Siblings were requested to come monthly for dietary counseling. Smoking cessation interventions used individual counseling previously carried out by the investigators. Smoking assessment included self-report and measures of carbon monoxide (CO) in expired air. Study physicians carried out pharmacologic interventions for blood pressure, lipids and lipoproteins. Diabetes treatment was through referral to the patient's private physician. Nurses provided oversight to NHWs.

Neighborhood health workers were trained and certified in taking blood pressure (BP), phlebotomy, and CO measurements at the Center for Health Promotion at Johns Hopkins, which had an NHW training program for blood pressure. Outcomes measures included changes in blood pressure, smoking behavior, and plasma concentrations of lipids and lipoproteins. Attention was paid to potential modifying factors such as demographic factors (e.g., education, socioeconomic status, income, occupation).

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Healthy Black siblings of individuals with premature coronary disease. Over 60% were women. Sibs were eligible if they were aged between 30 and 59 years with no known history of CAD, no chronic glucocorticosteroid therapy, no autoimmune disease, no current cancer therapy, and no immediate life-threatening comorbidity.

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1998-04; Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane Becker — Johns Hopkins University

REFERENCES:
- [Background] Becker DM, Tuggle MB, Prentice MF. Building a gateway to promote cardiovascular health research in African-American communities: lessons and findings from the field. Am J Med Sci. 2001 Nov;322(5):288-93. PMID 11721804
- [Background] Mora S, Yanek LR, Moy TF, Fallin MD, Becker LC, Becker DM. Interaction of body mass index and framingham risk score in predicting incident coronary disease in families. Circulation. 2005 Apr 19;111(15):1871-6. doi: 10.1161/01.CIR.0000161956.75255.7B. PMID 15837938
- [Background] Becker DM, Yanek LR, Johnson WR Jr, Garrett D, Moy TF, Reynolds SS, Blumenthal RS, Vaidya D, Becker LC. Impact of a community-based multiple risk factor intervention on cardiovascular risk in black families with a history of premature coronary disease. Circulation. 2005 Mar 15;111(10):1298-304. doi: 10.1161/01.CIR.0000157734.97351.B2. PMID 15769772
- [Background] Benton JL, Blumenthal RS, Becker DM, Yanek LR, Moy TF, Post W. Predictors of low-density lipoprotein particle size in a high-risk African-American population. Am J Cardiol. 2005 Jun 1;95(11):1320-3. doi: 10.1016/j.amjcard.2005.01.075. PMID 15904636